CLINICAL TRIAL: NCT07007936
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase IIa Trial to Evaluate the Efficacy and Safety of Oral SSS17 Capsules in the Treatment of Anemia Following Total Hip or Knee Arthroplasty
Brief Title: Phase IIa Trial of Oral SSS17 for Post-Arthroplasty Anemia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shenyang Sunshine Pharmaceutical Co., LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SSS17-202
Record Dates: First submitted 2025-05-29; First posted 2025-06-06 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Anemia; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
MeSH Terms: interventions — Floors and Floorcoverings

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSS17 (Experimental): The study employs a hybrid design with six dose levels: four fixed-dose parallel arms and two sequential dose-escalation cohort
  Interventions: Drug: SSS17 Capsule (6 Dose Levels); Drug: Placebo Drug
- placebo (Placebo Comparator)
  Interventions: Drug: SSS17 Capsule (6 Dose Levels); Drug: Placebo Drug

INTERVENTIONS:
Drug: SSS17 Capsule (6 Dose Levels) — Arm1 ： This dose-ranging study evaluates 6 dose levels of oral SSS17 capsules under two regimens: Once weekly、 Twice weekly
Drug: Placebo Drug — Arm2：placebo The placebo intervention was matched with the six dose levels of SSS17, with each dose level assigning participants in a ratio of 4:1 (SSS17 to placebo).

SUMMARY:
To assess the safety, tolerability, efficacy, and pharmacokinetic/pharmacodynamic (PK/PD) characteristics of orally administered SSS17 capsules in patients with postoperative anemia following elective total hip or knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent obtained

   -
2. Age 18-70 years (inclusive)

   -
3. Candidates for hip/knee arthroplasty

   -
4. No DVT on pre-op venous ultrasound

   -
5. Screening Hb 80-110 g/L (no transfusion indication) - 6. Commitment to effective contraception

Exclusion Criteria:

1. Hypersensitivity to the investigational product or any of its components
2. Any other condition causing chronic anemia
3. Coagulopathy or unstable anticoagulant dosing during screening
4. Any of the following laboratory abnormalities at screening:

   1. Serum albumin <35 g/L
   2. ALT or AST >3×ULN
5. Active infections or carrier status including:

   * Known HIV infection
   * Active syphilis
   * Active HBV infection (HBsAg-positive with HBV DNA >10³ copies/mL)
   * Active HCV infection (anti-HCV positive with detectable HCV RNA)
6. Acute joint injury with active trauma or infection at screening
7. Cognitive impairment or psychiatric disorders,current or history of epilepsy
8. Treatment with ESAs (erythropoiesis-stimulating agents) or HIF inhibitors within 30 days prior to dosing
9. History of severe thromboembolic events or hematopoietic disorders
10. Malignancy history
11. Severe cardiovascular diseases including:

    * Unstable coronary artery disease
    * Heart failure (NYHA Class III/IV)
    * Myocardial infarction/stroke 12 .Poorly controlled hypertension

13. Alcohol abuse 14.Pregnancy or lactation 15.Participation in other drug trials within 3 months prior to enrollment 16.Any other condition deemed by the Investigator to compromise subject safety or trial validity

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in hemoglobin | Day 8，Day 15，Day 29

SECONDARY OUTCOMES:
Proportion of subjects requiring transfusion and transfusion volume | Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided